CLINICAL TRIAL: NCT05815407
Title: The Expression Profiling of Serum miRNAs (106b-5p, 601, and 760) in Non-small Cell Lung Cancer Patients
Brief Title: Expressiona and Diagnostic Potential of miRNAs in NSCLC
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Collaborators: National Cancer Institute, Cairo University, Egypt (Unknown)
Responsible Party: Principal Investigator, Ahmed Elshafei, Professor Associate of Medical Biochemistry and Molecular Biology, Al-Azhar University
Other Study IDs: FOP AlAzharU
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC patients: Patients were diagnosed with NSCLC at any stage, then will be subdivided into Early stage, Lympho-node involvement stage and Distant metastatic stage
  Interventions: Other: No intervention
- Control subjects: Appearantly healthy age-matched individuals
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Its to explore the expression pattern, diagnostic and prognostic potentials of miRs (106b-5p, 601 and 760) in serum of NSCLC patients

DETAILED DESCRIPTION:
A retrospective observational study on NSCLC patients, to determine the serum expression levels if some miRNAs in NSCLC patients and to find if having proper diagnostic and prognostic values in early disease detection, and/or staging.

ELIGIBILITY:
Inclusion Criteria:

* First time and recently diagnosed NSCLC patient

Exclusion Criteria:

* Recurrent NSCLC
* Start of chemotherapy, radiotherapy or surgical intervention
* Previous treatment
* Cancer history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case-control
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Determination of the expression | By the end of the study (September 2022)
  Expression profiling of the selected miRNAs

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Al-Azhar University, Cairo, Egypt, Cairo, Egypt